CLINICAL TRIAL: NCT07097805
Title: Glycemic Improvement With Team, Technology, Education and Peer Resources in Type 1 Diabetes-GLITTER Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KYZ20240193
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; Comprehensive management
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T1D Patients (Other): All patients diagnosed with type 1 diabetes of all ages.
  Interventions: Behavioral: GLITTER comprehensive management

INTERVENTIONS:
Behavioral: GLITTER comprehensive management — The GLITTER comprehensive management represents a management approach that effectively combines multidisciplinary professional team care, diabetes technology empowerment, structured education steering, and peer support.

SUMMARY:
The GLITTER study is comprised of four key components: Team, Technology, Education, and Peer Resources. The aim of the GLITTER Study is to improve the metabolic control rate in patients with type 1 diabetes through a comprehensive management approach.

DETAILED DESCRIPTION:
Patients with type 1 diabetes (T1D) face significant glycemic fluctuations, posing substantial challenges in disease management. Current clinical evidence indicates that although interventions such as structured education programs, peer support, and novel diabetes technologies demonstrate positive outcomes when applied individually, the glycemic target attainment rate remains suboptimal, with fewer than 30% achieving this benchmark. To address this clinical dilemma, the investigators has proposed the GLITTER (Glycemic Improvement with Team, Technology, Education and Peer Resources in type 1 diabetes) study, which aims to establish a four-in-one integrated management model combining multidisciplinary collaborative teams, structured educational frameworks, peer support systems, and diabetes technologies. The research team comprises T1D-specialized physicians and diabetes educators. Structured education is delivered through dedicated T1D specialty clinics and by local clinicians. Technological support involves informing patients about access to continuous glucose monitors (CGM) and insulin pumps without mandating their use, while peer support is established through patient communication groups (volunteer matching mechanisms are not yet implemented). This GLITTER study seeks to achieve dual objectives: population-wide coverage and whole-disease-course management for individuals with T1D.

This is a multicenter, prospective, cohort study. This longitudinal investigation systematically collects multidimensional clinical datasets encompassing glycemic control parameters, pancreatic β-cell function, and complication risk profiles through regular follow-up visits. This study explores the metabolic control, psychological outcomes, and their associated influencing factors among patients with T1D.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 1 diabetes of all age groups, regardless of disease duration.

The diagnosis criteria for type 1 diabetes are met by fulfilling any one point from the first two criteria plus any one point from the third criterion.

1. Clinically diagnosed as Type 1 Diabetes by a specialist physician.
2. Meet any one of the following criteria:

   A. Age of onset <15 years B. No obesity at the time of onset C. diabetic ketoacidosis onset D. Maximum random C-peptide <200 pmol/L
3. Meet any one of the following criteria:

A. Initiation and continuation of insulin therapy after diagnosis (excluding pancreas or islet transplantation) B. Positive for islet cell antibodies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Trough study completion, an average of 1 year
  The primary outcome is the Change in Glycated Hemoglobin A1C (HbA1c). HbA1c is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.

SECONDARY OUTCOMES:
Percentage of patients using continuous glucose monitors | Trough study completion, an average of 1 year
  The percentage of participants who initiate and maintain active use of a continuous glucose monitor (CGM) trough study completion. Active use is defined as wearing the CGM sensor and having recorded glucose data available. Confirmation will be based on CGM device data download or patient self-reported daily wear logs verified by research staff or electronic adherence monitoring from the CGM cloud platform.
Percentage of patients using insulin pump | Trough study completion, an average of 1 year
  Proportion of enrolled patients maintaining active insulin pump use during follow-up, defined as consistent pump utilization confirmed by either:
  1. Device data download demonstrating functional use; or
  2. Clinician-verified patient logbook records with corroborating evidence.
Diabetes-related complications | Trough study completion, an average of 1 year
  Diabetes-related complications encompass microvascular disorders (diabetic retinopathy, nephropathy, neuropathy), macrovascular complications (coronary artery disease, cerebrovascular disease, peripheral arterial disease), neuropathic complications (peripheral neuropathy, autonomic neuropathy), diabetic foot syndrome, and acute metabolic events (severe hypoglycemia, ketoacidosis, hyperosmolar hyperglycemic state, diabetic lactic acidosis).
Urine Albumin-to-Creatinine Ratio | Trough study completion, an average of 1 year
  Normal: <30 mg/g；Microalbuminuria: 30-300 mg/g；Macroalbuminuria: >300 mg/g
Change in titer of autoantibodies | Trough study completion, an average of 1 year
  Islet autoantibodies represent serological markers of autoimmune destruction targeting pancreatic β-cell antigens, serving as pivotal biomarkers for T1D pathogenesis.
Change in C-peptide | Trough study completion, an average of 1 year
  C-peptide are measured before and 2-hour after a mixed meal tolerance test at each follow-up of this study.
Change in blood glucose | Trough study completion, an average of 1 year
  Blood glucose are measured before and 2-hour after a mixed meal tolerance test at each follow-up of this study.
Systolic blood pressure | Trough study completion, an average of 1 year
  Systolic blood pressure
Diastolic blood pressure | Trough study completion, an average of 1 year
  Diastolic blood pressure
Change in lipid profiles | Trough study completion, an average of 1 year
  Including triglyceride, total cholesterol, HDL-cholesterol and LDL-cholesterol
Self-Management of Type 1 Diabetes for Chinese Adults | Trough study completion, an average of 1 year
  The Self-Management of Type 1 Diabetes for Chinese Adults (SMOD-CA) scale is a validated instrument specifically designed to assess the self-management behaviors and capabilities of adults with type 1 diabetes in the Chinese population. The SMOD-CA consists of 30 items. Responses are rated on a five-point scale, with higher scores indicating better self-management ability. The total score ranges from 0 to 120.
23-item Chinese Version of Self-Report Measure of Self-Management of Type 1 Diabetes for Adolescents | Trough study completion, an average of 1 year
  The 23-item Chinese Version of Self-Report Measure of Self-Management of Type 1 Diabetes for Adolescents (C-SMOD-A-23) is a validated and simplified instrument designed to assess the self-management behaviors and capabilities of adolescents with type 1 diabetes.
Chinese version of the Diabetes Quality of Life for Youth Scale Short Form | Trough study completion, an average of 1 year
  The Chinese version of the Diabetes Quality of Life for Youth Scale Short Form (C-DQOLY-SF) is a psychometrically tested instrument designed to assess the quality of life in adolescents with type 1 diabetes. The scale consists of 25 items that measure various aspects of life satisfaction, diabetes impact, and diabetes-related worry.
Athens Insomnia Scale | Trough study completion, an average of 1 year
  The Athens Insomnia Scale (AIS) is a self-assessment tool used to evaluate the presence and severity of insomnia symptoms. The total score provides a quantitative measure of insomnia severity, with higher scores indicating more significant sleep disturbances.
Depression Self-Rating Scale for Children | Trough study completion, an average of 1 year
  The Depression Self-Rating Scale for Children (DSRSC) is a standardized psychological assessment tool designed to measure depressive symptoms in children and adolescents. This self-report inventory allows young individuals to rate the frequency and severity of various depressive feelings and behaviors they may be experiencing.
Diagnosis and measurement of the severity of depression: Patient Health Questionnaire | Trough study completion, an average of 1 year
  The Patient Health Questionnaire (PHQ-9) will be used to assess depressive symptoms, including suicidal ideation, over the last two weeks (9 questions). Items are scored 0-3, resulting in a total score of 0-27. Higher scores indicate more symptoms of depression.
Generalized Anxiety Disorder 7-item scale | Trough study completion, an average of 1 year
  The Generalized Anxiety Disorder 7-item scale (GAD-7) consists of seven items. Each item asks respondents to rate how often they have been bothered by specific anxiety-related symptoms over the past two weeks.
WHO-5 Well-Being Index | Trough study completion, an average of 1 year
  The WHO-5 Well-Being Index (WHO-5) is a brief, self-report questionnaire designed to assess subjective well-being. The WHO-5 consists of five simple and straightforward items. Each item is rated on a 6-point Likert scale, ranging from 0 (not present) to 5 (constantly present). The total score is calculated by summing the responses to all five items, resulting in a score that ranges from 0 to 25. Higher scores indicate better well-being.
Mini-EAT | Trough study completion, an average of 1 year
  The Mini-Eating Assessment Tool, is a brief dietary assessment scale designed to evaluate the quality of an individual's diet. It is a concise tool that aims to provide a quick yet effective measure of dietary habits and nutrition intake.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Department of Endocrinology and Metabolism, Peking University People's Hospital, Beijing, Beijing Municipality
  - Department of Endocrinology, Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Department of Endocrinology and Metabolism, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Department of Endocrinology, Shenzhen Second People's Hospital, The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong
  - Endocrinology and Metabolism Center, The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan
  - Institute of Metabolism and Endocrinology, Second Xiangya Hospital of Centra South University, Changsha, Hunan
  - Department of Endocrinology, The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Department of Endocrinology and Metabolism, Institute of Endocrinology, The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Department of Endocrinology and Metabolism, Laboratory of Diabetes and metabolism research, West China Hospital, Sichuan University, Chengdu, Sichuan
  - Department of Endocrinology, Children's Hospital of Zhejiang University School of Medicine, National Clinical Research Center for Child Health, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No